CLINICAL TRIAL: NCT06437847
Title: Assessment of the Need to Use Short Cognitive Tests for French General Practitioners/Family Doctors
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN632024/CHUSTE
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Disorder
Keywords: Cognitive evaluation; Short Test; General Practitioners; Codex, Training; Formation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire assessing the use of cognitive tests.

SUMMARY:
The prevalence of cognitive disorders is constantly increasing, with 1.2 million patients affected in France in 2016. Dementia is currently the seventh leading cause of death. In the absence of available treatment, systematic screening is not recommended. However, cognitive evaluation is recommended to maintain a level of autonomy for the patient at home. Targeted screening is the responsibility of the general practitioner. The latest recommendations from the HAS (2011) highlight the use of the MMSE as a first-line approach, there are no recommendations regarding short tests. Early cognitive assessment is limited by the time required to perform the tests and the knowledge about the available tools. The Codex is a short test, its sensitivity (92%) and specificity (85%) place it among the most discriminatory scores. It is underutilized in France. The objective of this thesis is to assess the training needs of general practitioners in short tests.

ELIGIBILITY:
Inclusion Criteria:

* General practitioners of the AURA Region, in activity, university supervisor or not, trained or not trained in geriatrics.

Exclusion Criteria:

* General practitioners with exclusive practices in pediatrics, gynecology, aesthetics, rehabilitation, and homeopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General practitioners of the AURA Region will be included.
Sampling Method: Non-Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Quantitative questionnaire 1 | Month : 1, 3, 6
  Assessment of the need to use short cognitive tests

SECONDARY OUTCOMES:
Quantitative questionnaire 2 | Month : 1, 3, 6
  Assessment of the expectation regarding a project of training general practitioners to use the Codex tool (Sum = 4 or 5: = CODEX normal ; Sum = 0, 1, 2 or 3 = CODEX abnormal)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No